CLINICAL TRIAL: NCT06770894
Title: A Randomized, Double Blind Placebo Controlled Clinical Trial to Assess the Efficacy and Safety of Sitagliptin on Bone Measures in Women Affected by Type 2 Diabetes. a Gender-oriented Approach to Address a Gender-specific Frailty: the SLowDOWN (SitagLiptin in Diabetes for Osteoporosis in WomeN) Study.
Brief Title: DPP4-Inhibitors and Bone Metabolism in Diabetes
Acronym: SlowDOWN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Policlinico Umberto I (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Principal Investigator, Maria Gisella Cavallo, Professor, Azienda Policlinico Umberto I
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AIFA-2016-02364864; 2018-000859-40 (EudraCT Number)
Record Dates: First submitted 2025-01-02; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Osteoporosis; Bone Loss, Postmenopausal; Diabetes Mellitus Type 2
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal; Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active treatment (Experimental): Sitagliptin 100 mg, 1 tablet per day
  Interventions: Drug: Sitagliptin 100 mg
- Placebo (Placebo Comparator): Placebo tablets, provided in identical blisters
  Interventions: Drug: Placebo Tablets

INTERVENTIONS:
Drug: Sitagliptin 100 mg — The study population will be randomly allocated in either intervention or placebo arm (1:1). Treatment (sitagliptin 100 mg) and placebo will be provide in identical packages by an experienced independent pharmacist. The recommended intake is one tablet a day, equivalent to sitagliptin 100 mg in the active-treated group, for the duration of the study (52 weeks)
  Arms: Active treatment
Drug: Placebo Tablets — Placebo tablets 1 a day, provided in identical blisters.
  Arms: Placebo

SUMMARY:
Background Bone frailty and fractures are common conditions in patients with type 2 diabetes (T2D) and represent a major cause of morbidity and hospitalization in this population. In women, the postmenopausal period is well known to dramatically impact bone mineralization and metabolism, leading to a higher risk of bone fractures. Additionally, hyperglycemia, oxidative stress, and advanced glycation end-products accumulation, as occur in diabetes, negatively impact bone quality. Thus, the coexistence of T2D in postmenopausal women represents a detrimental condition highly increasing the risk of bone fractures and hospitalization.

Dipeptidyl peptidase 4 inhibitors (DPP4-Is) are a promising class of antidiabetic agents with protective effects on bone in experimental conditions. In vivo, higher DPP4 activity correlates with lower bone mineral density (BMD) in women, and DPP4-Is treatment was associated with favorable bone outcomes in the only meta-analysis available on subjects with T2D. However, whether chronic DPP4-I treatment is capable of improving bone outcomes in women affected by T2D has not been explored yet in the context of a specifically designed clinical trial.

Objectives This study is a superiority, double-blinded, randomized, placebo-controlled clinical trial aiming to investigate the safety and efficacy of 52-week sitagliptin 100 mg therapy in improving bone outcomes in women affected by T2D.

Methods For this purpose, the investigators aim to recruit 132 female patients aged ≥18 years with a diagnosis of T2D, BMI between 20-40 kg/m², body weight ≤120 kg, and HbA1c between 6.5 and 7.5%, undergoing treatment with metformin in monotherapy at a stable dose for ≥12 weeks prior to recruitment. The enrolment setting is the Diabetes Outpatients' Clinics, Policlinico Umberto I, Sapienza University of Rome. Screening will be performed among all patients referred to these clinics for diabetes care. Both recruitment and intervention are anticipated to take place over a 36-month period.

Primary outcome measures are: (1) changes in bone mineral density (BMD), estimated by dual-energy x-ray absorptiometry (DXA) for the lumbar spine and femoral neck, and (2) changes in markers of bone formation/resorption from baseline to the end of treatment (week 52). Secondary endpoints are: (I) evaluation of the association between circulating DPP4 activity and serum markers of bone metabolism at baseline and after 24- and 52-week sitagliptin treatment; (II) determination of whether circulating DPP4 activity is associated with impaired vitamin D availability; and (III) investigation of the relationship between DPP4 activity and systemic markers of inflammation throughout the study.

Expected Results Both T2D and osteoporosis are widespread conditions with a strong impact on life expectancy, quality of life, and healthcare costs. It has been estimated that a quarter of all women will suffer from osteoporosis after menopause, with a 30-40% risk of osteoporotic fractures in their lifetime-much higher than the overall risk of breast, uterine, and ovarian cancer. In Italy, osteoporosis accounts for 500 million Euros in hospitalization costs and is associated with high rates of disability with profound social and psychological impacts.

On the other hand, DPP4-Is represent a widespread treatment for T2D, capable of providing adequate glycemic control with a very low risk of hypoglycemia and serious adverse events. Therefore, this study will provide novel and original evidence on the effects of DPP4-Is on bone health in the context of a specifically designed randomized clinical trial. It will address specific frailties in women, such as osteoporosis and fractures, the risk of which is further increased in the presence of diabetes. The demonstration of favorable effects of chronic DPP4-I treatment on bone metabolism may guide clinicians among the large number of therapeutic options for diabetes care, with immediate implications for a multi-approach diabetes treatment strategy.

DETAILED DESCRIPTION:
This study is a superiority, double-blinded, randomized, placebo-controlled clinical trial designed to investigate the safety and efficacy of 52-week sitagliptin 100 mg therapy in improving bone outcomes in women affected by type 2 diabetes.

In particular, the primary objective of this study is:

To test the superiority of sitagliptin 100 mg in addition to metformin versus placebo with metformin in improving bone mineral density from baseline to the end of treatment (week 52), as estimated by DXA on the lumbar spine and femoral neck.

Secondary endpoints are:

Evaluation of the association between circulating DPP4 activity and serum markers of bone metabolism at baseline and after 24- and 52-week sitagliptin supplementation.

Determination of whether circulating DPP4 activity is associated with impaired vitamin D availability and whether chronic DPP4 inhibition induces changes in serum vitamin D levels after treatment.

Examination of the relationship between DPP4 activity and systemic markers of inflammation, which are closely related to impaired glucose metabolism, at baseline and after 24- and 52-week sitagliptin supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects ≥ 18 years
* Diagnosis of Type 2 Diabetes according to American Diabetes Association 2009 criteria
* Body mass index (BMI) between 20-40 kg/m2
* Body weight ≤ 120 kg (due to limitations imposed by DXA equipment);
* HbA1c < 7.5%
* Treatment with metformin in monotherapy at a stable dose for ≥12 weeks prior to enrolment
* Women not of childbearing potential may participate and include those who are:

I) infertile due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation), congenital anomaly such as Mullerian agenisis; or II) postmenopausal - defined as either

1. A woman 50 to 54 years of age (inclusive) with an intact uterus, not hormone therapy who has had either

   1. cessation of menses for at least 1 years or
   2. at least 6 months of spontaneous amenorrhea with a follicle-stimulating hormone > 40 mIU/mL; or
2. a woman 55 or holder not on hormone therapy, who has had at least 6 months of spontaneous amenorrhea; or
3. a woman at least 55 years of age with a diagnosis of menopause prior to starting hormone replacement therapy - Women of childbearing potential participating: I) cannot be pregnant or intend to become pregnant II) cannot be breastfeeding III) must remain abstinent or use 1 highly effective method of contraception or combination of 2 effective methods of contraception for the entirety of the study IV) test negative for pregnancy at the time of screening

Exclusion Criteria:

* Treatments known to significantly influence bone metabolism (e.g. bisphosphonates, calcitonin, corticosteroids or hormone replacement therapy)
* Osteomalacia
* Paget.s disease
* Hyperparathyroidism
* Hyperthyroidism
* Chronic liver failure/cirrhosis
* Kidney failure
* Current or history of therapy with antidiabetic agents other than metformin
* Pregnancy/lactation, childbearing potential women who do not give their consent to remain abstinent or use 1 highly effective method of contraception or combination of 2 effective methods of contraception for the entirety of the study
* Pregnancy/lactation
* Substance abuse, clinically significant depression or current psychiatric care
* Refuse or are unable to give informed consent to participate in the study Subjects taking vitamin D and/or calcium supplements at enrolment will be instructed to continue this therapy keeping the doses unchanged throughout the entire study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 132 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Change in Bone Mineral Density (BMD) at Lumbar Spine and femoral neck (g/cm²) | Baseline to 52 weeks
  To assess the change in bone mineral density at the lumbar spine and femoral neck from baseline to the end of treatment (week 52), estimated by dual-energy X-ray absorptiometry (DXA).
  Unit of Measure: g/cm²

SECONDARY OUTCOMES:
Correlation Between Circulating DPP4 Activity and Serum Markers of Bone Metabolism and Inflammation | baseline, 24 weeks and 52 weeks
  To evaluate the correlation between circulating DPP4 activity (nmol/min/mL) and serum markers of bone metabolism (OPG, OPN, OC, CTX; measured in ng/mL), inflammation (TNFa, ILs; measured in pg/mL) and 25(OH)vitamin D levels (ng/mL) at the baseline and after 24 and 52 weeks of sitagliptin supplementation.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Policlinico Umberto I, University La Sapienza, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
De-identified, aggregated raw data may be shared upon reasonable request, subject to review and approval by the Principal Investigator (PI). Requests must be justified with a clear scientific purpose and comply with applicable ethical and regulatory standards.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Barchetta I, Filardi T, Dule S, Cimini FA, Sentinelli F, Romagnoli E, Passarella G, Bleve E, Oldani A, Venditti V, Anastasi E, Gandini O, Napoli N, Nicolucci A, Lenzi A, Baroni MG, Morano S, Cavallo MG; SlowDOWN Study Network. Effect of sitagliptin vs. placebo on bone mineralization in women with type 2 diabetes: the SLowDOWN (SitagLiptin in Diabetes for Osteoporosis in WomeN) randomized clinical trial. BMC Med. 2025 Oct 14;23(1):562. doi: 10.1186/s12916-025-04363-w. PMID 41088165